CLINICAL TRIAL: NCT03731286
Title: A Double-Blind Randomized, Double-dummy, Placebo-controlled, Parallel-Group Study of the Long-term Safety and Efficacy of EnXtra (E-AG-01) in Healthy Adults
Brief Title: A Long-term Safety and Efficacy of EnXtra (E-AG-01) in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: EB/180401/ENXTRA/EVRG
Record Dates: First submitted 2018-10-29; First posted 2018-11-06 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2018-10

CONDITIONS: Caffeine Dependence
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Alpinia galanga (Active Comparator): EnXtra: 2 capsules to be taken twice daily after breakfast and evening.
  Interventions: Dietary Supplement: Alpinia Galanga
- Composite (Alpinia galanga + Caffeine) (Active Comparator): Composite: 2 capsules to be taken twice daily after breakfast and evening.
  Interventions: Dietary Supplement: Alpinia Galanga
- Placebo (Placebo Comparator): Microcellulose crystalline: 2 capsules to be taken twice daily after breakfast and evening.
  Interventions: Dietary Supplement: Microcellulose crystalline

INTERVENTIONS:
Dietary Supplement: Alpinia Galanga — 2 capsules
  Arms: Alpinia galanga
Dietary Supplement: Alpinia Galanga — 2 capsules
  Other Names: Caffeine
  Arms: Composite (Alpinia galanga + Caffeine)
Dietary Supplement: Microcellulose crystalline — 2 capsules
  Arms: Placebo

SUMMARY:
The present study has been proposed to investigate the long-term safety and efficacy of EnXtra in healthy adults habituated to caffeine.

ELIGIBILITY:
Inclusion Criteria:

1. History of regular caffeine consumption.
2. Body mass index (BMI) of ≥18.5 and <25.00 kg/m2.
3. Fasting blood glucose < 126 mg/dl
4. Participants who are willing to complete all study procedures including study-related questionnaires and comply with study requirements.
5. Participants who are willing to abstain from use of any nutritional supplement and herbal preparation 48 hrs prior to study visit.

Exclusion Criteria:

1. Participants unable to abstain from caffeine-containing products for 12 hours prior to the site visit.
2. Known cases of type II Diabetes Mellitus.
3. Participants with uncontrolled hypertension (≥140/90 mm Hg), with or without anti-hypertensive medication.
4. Participants suffering from primary or secondary insomnia with/ without active treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-23 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Change in ECG from baseline to end of the treatment. | 84 Days
  ECG parameters including PR interval, QRS duration, QT interval and RR interval will be evaluated from baseline and end of the treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Vedic Lifesciences Pvt. Ltd, Mumbai, Opp Infinity Mall, India